CLINICAL TRIAL: NCT01562886
Title: A Phase I Pharmacokinetic Study to Assess the Cerebrospinal-fluid (CSF) Exposure of Rilpivirine in HIV-infected Subjects Switching From TDF/FTC/Nevirapine to TDF/FTC/Rilpivirine
Brief Title: The Rilpivirine Cerebrospinal-fluid (CSF) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 278_CSF; 2011-004026-98 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-05

CONDITIONS: HIV
Keywords: Rilpivirine CSF pharmacokinetics
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rilpivirine and Truvada (Experimental): TDF/FTC (Truvada™) one tablet once plus Rilpivirine 25 mg daily
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Rilpivirine — Rilpivirine 26mg
  Other Names: Edurant

SUMMARY:
This is a phase I pharmacokinetic study of HIV positive patients stable on antiretroviral therapy who will switch treatment when enrolled from nevirapine to rilpivirine. On day 60 of the study the participants will attend clinic where they will have blood collected followed by a lumbar puncture where cerebrospinal fluid will be collected to measure drug concentration. The participants will then restart their original regime with nevirapine.

DETAILED DESCRIPTION:
To investigate the following parameters in HIV-infected patients switching antiretroviral therapy from TDF/FTC/nevirapine to TDF/FTC/rilpivirine for 60 days:

* CSF exposure and CSF : plasma ratio of rilpivirine
* Safety and tolerability of switching antiretroviral therapy from TDF/FTC/nevirapine to TDF/FTC/rilpivirine
* Changes in cerebral metabolites measured via 1-H MRS after switching antiretroviral therapy to TDF/FTC/rilpivirine
* Seminal fluid exposure of rilpivirine

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males subjects
* signed informed consent
* willing to switch therapy as per study protocol
* no previous exposure to rilpivirine
* plasma HIV RNA < 50 copies/mL at screening and on at least one other occasion over the last 3 months
* currently receiving a stable antiretroviral regimen comprising of TDF/FTC with nevirapine with nevirapine dosed either 200 mg twice daily or 400 mg once daily with no antiretroviral drug switches for at least 3 months
* no clinically-significant resistance documented on any prior HIV-1 genotypic resistance testing
* subjects in good health upon medical history, physical exam, and laboratory testing
* BMI above or equal to 18 and below 32
* Male subjects who are heterosexually active must use two forms of barrier contraception (e.g., condom and diaphragm) during heterosexual intercourse, from screening through completion of the study.
* Have local screening laboratory results (haematology and chemistry that fall within the normal range of the central laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance
* No contraindications to having a lumbar puncture examination found on MRI of the brain

Exclusion Criteria:

* current alcohol abuse or drug dependence
* positive urine drug of abuse screening
* active opportunistic infection or significant co-morbidities
* current disallowed concomitant medication (as listed in section 4.1.3)
* contraindication to MR examination or lumbar puncture examination
* recent head injury (in last 30 days) or chronic ongoing neurological diseases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MBChB MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rilpivirine and Truvada
Started | 14
Completed | 13
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rilpivirine and Truvada
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13
Rilpivirine CSF concentration [Geometric Mean (Full Range); unit: ng/mL] | 0.8 [0.54 to 1.57]

OUTCOME MEASURES:

1. Primary Outcome: CSF:Plasma Ratio of Rilpivirine Levels
Description: The levels of rilpivirine will be measured in the cerebral spinal fluid and plasma after 60 days of exposure
Time Frame: Day 60
Measure: Geometric Mean (95% Confidence Interval); unit: ratio expressed as a percentage
Groups:
- Rilpivirine and Truvada: TDF/FTC (Truvada™) one tablet once plus Rilpivirine 25 mg daily
  Rilpivirine: Rilpivirine 25mg
Arm/Group | Rilpivirine and Truvada
Number analyzed (Participants) | 13
ratio expressed as a percentage | 1.4 [1.2 to 1.6]

2. Secondary Outcome: Number of Subjects With HIV Viral Load Above 50 Copies Per mL
Description: Plasma viral load will be measured at all study visits to assess if viral load is above the lower limit of detection (50 copies mL)
Time Frame: Day 3,14, 28, 60, 80-100
Measure: Number; unit: participants
Arm/Group | Rilpivirine and Truvada
Number analyzed (Participants) | 13
participants | 2

ADVERSE EVENTS:
Time Frame: Duration of the study
Arm/Group | Rilpivirine and Truvada
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rilpivirine and Truvada (N=13)
Insomnia (Nervous system disorders) | 3 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No